CLINICAL TRIAL: NCT03860389
Title: The Effects of a School Based Exercise Programme on Behaviour and Anxiety in Children With ASD
Brief Title: The Effects of Exercise in Anxiety in Children With ASD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Technology, Carlow (Other)
Collaborators: University of Reading (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASD1
Record Dates: First submitted 2019-02-12; First posted 2019-03-01 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Autism Spectrum Disorder; Anxiety; Behavior
Keywords: Autism; Anxiety; Exercise; Behaviour
MeSH Terms: conditions — Autism Spectrum Disorder; Anxiety Disorders; Behavior; Autistic Disorder; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise effects on anxiety (Experimental): An exercise programme will be administered 3 times a week for up to an 16 week period of time in a school setting. Each exercise class will last 60 minutes. The exercise classes will involve aspects of fundamental movement skills and will be fun for the students to participate in.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — An exercise programme will be delivered in the school for a period of up to 16 weeks. Exercise classes will take place 3 times a week and will be of 60 minutes duration.

SUMMARY:
This study will examine the effects of a school based exercise programme on anxiety and behaviour levels in children with autism.

DETAILED DESCRIPTION:
This study will examine the effects of a school based exercise programme on anxiety and behaviour levels in children with autism. Local special autism schools and primary and secondary schools with specialised classes for children with autism will be approached to participate in the project. The age profile of the children will be 4-18 yrs of age and they will have mild-severe levels of autism. The exercise programme will delivered 3 times per week in the schools over periods of 8-16 weeks dependent on the severity of autism within the children.

Questionnaires will be given to the parents and teachers of the children at the beginning and at the end of the programme to assess changes in anxiety levels and behaviour as a result of the exercise programme.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of autism spectrum disorder

Exclusion Criteria:

* Any medical condition which excludes the child from partaking in exercise

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-01-07 (Actual); Primary Completion 2019-06-24 (Estimated); Study Completion 2019-12-16 (Estimated)

PRIMARY OUTCOMES:
Anxiety | Change from baseline at Week 8 and Week 16
  Changes in anxiety levels of the children will be assessed using the Anxiety Scale for Children -ASD.
Behaviour | Change from baseline at Week 8 and Week 16
  Changes in the behaviour of the children will be assessed using the Nisingor Child Behaviour Rating Form

SECONDARY OUTCOMES:
Fitness level | Change from baseline at Week 8 and Week 16
  The modified Eurofit test will be used to assess the fitness levels of children

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Kinsella, PhD, Principal Investigator — IT Carlow
Locations (1):
- Sharon Kinsella, Carlow, Co. Carlow, Ireland

IPD SHARING:
Plan to Share IPD: Undecided